CLINICAL TRIAL: NCT00694707
Title: Evaluation of the Safety and Efficacy of RGH-188 in the Acute Exacerbation of Schizophrenia
Brief Title: Safety and Efficacy of Cariprazine (RGH-188) in the Acute Exacerbation of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-16; NCT00892528 (obsolete NCT alias)
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo orally once a day for 6 weeks.
  Interventions: Drug: Placebo
- Cariprazine 1.5 mg (Experimental): Participants received cariprazine 1.5 mg orally once a day for 6 weeks.
  Interventions: Drug: Cariprazine
- Cariprazine 3.0 mg (Experimental): Participants received cariprazine 3.0 mg orally once a day for 6 weeks.
  Interventions: Drug: Cariprazine
- Cariprazine 4.5 mg (Experimental): Participants received cariprazine 4.5 mg orally once a day for 6 weeks.
  Interventions: Drug: Cariprazine
- Risperidone 4.0 mg (Active Comparator): Participants received risperidone 4.0 mg orally once a day for 6 weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Placebo — Placebo was supplied in capsules.
  Arms: Placebo
Drug: Cariprazine — Cariprazine was supplied in capsules
  Other Names: RGH-188
  Arms: Cariprazine 1.5 mg; Cariprazine 3.0 mg; Cariprazine 4.5 mg
Drug: Risperidone — Risperidone was supplied in capsules
  Other Names: Risperdal
  Arms: Risperidone 4.0 mg

SUMMARY:
This is a study to evaluate the safety, efficacy, and tolerability of cariprazine (RGH-188) relative to placebo in adult patients (18-60 years of age) with acute exacerbation of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 60 years of age.
* Meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for schizophrenia (paranoid type, disorganized type, catatonic type, or undifferentiated type) based on a Structured Clinical Interview for DSM-IV (SCID).
* Total Positive and Negative Syndrome Scale (PANSS) score ≥ 80 and ≤ 120.
* Diagnosis of schizophrenia for at least 1 year.

Exclusion Criteria:

* Abnormalities on physical examination or abnormal vital signs, electrocardiogram, or clinical laboratory values.
* First episode of psychosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 732 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2009-08-31 (Actual); Study Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Durgam, MD, Study Director — Forest Laboratories
Locations (55):
- United States (17):
  - Forest Investigative Site, Costa Mesa, California
  - Forest Investigative Site, Long Beach, California
  - Forest Investigative Site, Oceanside, California
  - Forest Investigative Site, Paramount, California
  - Forest Investigative Site, Riverside, California
  - Forest Investigative Site, Washington D.C., District of Columbia
  - Forest Investigative Site, Bradenton, Florida
  - Forest Investigative Site, Kissimmee, Florida
  - Forest Investigative Site, Lake Charles, Louisiana
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, Flowood, Mississippi
  - Forest Investigative Site, Bridgeton, Missouri
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Charleston, South Carolina
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Houston, Texas
  - Forest Investigative Site, Irving, Texas
- India (12):
  - Forest Investigative Site, Vijaywada, ANDH PRAD
  - Forest Investigative Site, Visakhapatnam, Andh Prad
  - Forest Investigative Site, Ahmedabad, Gujarat
  - Forest Investigative Site, Bangalore, Karna
  - Forest Investigative Site, Mangalore, Karna
  - Forest Investigative Site, Manipal, Karna
  - Forest Investigative Site, Mysore, Karna
  - Forest Investigative Site, Pune, Mahara
  - Forest Investigative Site, Jaipur, Rajasthan
  - Forest Investigative Site, Chennai, Tamil Nadu
  - Forest Investigative Site, Tirupati, Tamil Nadu
  - Forest Investigative Site, Kanpur, Uttar Prad
- Malaysia (5):
  - Forest Investigative Site, Johor Bahru, Johor
  - Forest Investigative Site, Kota Bharu, Kelantan
  - Forest Investigative Site, Lembah Pantai, Kuala Lumpur
  - Forest Investigative Site, Ipoh, Perak
  - Forest Investigative Site, Ulu Kinta, Perak
- Russia (11):
  - Forest Investigative Site, Arkhangelsk
  - Forest Investigative Site, Gatchina
  - Forest Investigative Site, Kazan'
  - Forest Investigative Site 1, Moscow
  - Forest Investigative Site 2, Moscow
  - Forest Investigative Site, Moscow
  - Forest Investigative Site, Nizhny Novgorod
  - Forest Investigative Site, Saint Petersburg
  - Forest Investigative Site 2, Saint Petersburg
  - Forest Investigative Site1, Saint Petersburg
  - Forest Investigative Site, Samara
- Ukraine (10):
  - Forest Investigative Site, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Forest Investigative Site, Donetsk, Donetsk Oblast
  - Forest Investigative Site, Kharkiv, Kharkivs’ka Oblast’
  - Forest Investigative Site, Hlevakha, Kyiv Oblast
  - Forest Investigative Site, Kyiv, Kyiv Oblast
  - Forest Investigative Site, Odesa, Odesa Oblast
  - Forest Investigative Site, Ternopil, Ternopil Oblast
  - Forest Investigative Site, Chernihiv
  - Forest Investigative Site, Kherson, Vil. Stepanivka
  - Forest Investigative Site, Kiev

REFERENCES:
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Marder S, Fleischhacker WW, Earley W, Lu K, Zhong Y, Nemeth G, Laszlovszky I, Szalai E, Durgam S. Efficacy of cariprazine across symptom domains in patients with acute exacerbation of schizophrenia: Pooled analyses from 3 phase II/III studies. Eur Neuropsychopharmacol. 2019 Jan;29(1):127-136. doi: 10.1016/j.euroneuro.2018.10.008. Epub 2018 Nov 20. PMID 30470662
- [Derived] Earley W, Durgam S, Lu K, Laszlovszky I, Debelle M, Kane JM. Safety and tolerability of cariprazine in patients with acute exacerbation of schizophrenia: a pooled analysis of four phase II/III randomized, double-blind, placebo-controlled studies. Int Clin Psychopharmacol. 2017 Nov;32(6):319-328. doi: 10.1097/YIC.0000000000000187. PMID 28692485
- [Derived] Citrome L, Durgam S, Lu K, Ferguson P, Laszlovszky I. The effect of cariprazine on hostility associated with schizophrenia: post hoc analyses from 3 randomized controlled trials. J Clin Psychiatry. 2016 Jan;77(1):109-15. doi: 10.4088/JCP.15m10192. PMID 26845266
- [Derived] Durgam S, Starace A, Li D, Migliore R, Ruth A, Nemeth G, Laszlovszky I. An evaluation of the safety and efficacy of cariprazine in patients with acute exacerbation of schizophrenia: a phase II, randomized clinical trial. Schizophr Res. 2014 Feb;152(2-3):450-7. doi: 10.1016/j.schres.2013.11.041. Epub 2014 Jan 10. PMID 24412468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Cariprazine 4.5 mg | Risperidone 4.0 mg
Started | 151 | 145 | 147 | 148 | 141
Completed | 79 | 90 | 96 | 98 | 101
Not Completed | 72 | 55 | 51 | 50 | 40
Not completed — Did Not Receive Treatment | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 22 | 14 | 8 | 12 | 13
Not completed — Insufficient Therapeutic Response | 33 | 18 | 17 | 15 | 10
Not completed — Protocol Violation | 1 | 2 | 1 | 3 | 1
Not completed — Withdrawal of Consent | 14 | 18 | 22 | 16 | 15
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0
Not completed — Jeopardizing Parole Status | 1 | 0 | 0 | 0 | 0
Not completed — Death in the Family | 1 | 0 | 0 | 0 | 0
Not completed — Arrest by Police | 0 | 1 | 0 | 0 | 0
Not completed — Administrative Reasons | 0 | 1 | 0 | 2 | 0
Not completed — Notification of Past Head Injury | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized participants who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Cariprazine 4.5 mg | Risperidone 4.0 mg | Total
Number analyzed (Participants) | 151 | 145 | 146 | 147 | 140 | 729
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.8) | 36.8 (9.6) | 37.1 (10.4) | 35.8 (10.8) | 36.5 (11.1) | 36.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 39 | 44 | 42 | 227
  Male | 101 | 93 | 107 | 103 | 98 | 502
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 2 | 4 | 5 | 24
  Not Hispanic or Latino | 145 | 138 | 144 | 143 | 135 | 705
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 0 | 3
  Asian | 36 | 34 | 37 | 39 | 37 | 183
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 34 | 32 | 38 | 32 | 35 | 171
  White | 80 | 77 | 71 | 75 | 67 | 370
  More than one race | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 74.4 (18.6) | 71.7 (17.7) | 74.8 (16.3) | 72.4 (16.6) | 75.1 (18.2) | 73.7 (17.5)
Height [Mean (Standard Deviation); unit: cm] | 170.8 (11.2) | 169.0 (10.5) | 170.7 (10.3) | 170.3 (10.4) | 170.0 (10.5) | 170.2 (10.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (4.5) | 24.9 (4.9) | 25.6 (4.6) | 24.8 (4.2) | 25.8 (4.8) | 25.2 (4.6)
Waist circumference [Mean (Standard Deviation); unit: cm] | 86.7 (12.9) | 85.2 (13.1) | 87.6 (12.6) | 85.8 (12.7) | 88.0 (13.0) | 86.7 (12.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item rating scale that assesses the positive and negative symptoms of individuals with schizophrenia. Responses to the 30 items are based on a structured clinical interview with the patient and on supporting clinical information obtained from family, hospital staff, or other reliable informants. Of the 30 psychiatric parameters measured by the scale, 7 assess positive symptoms (eg, delusions, grandiosity); 7 assess negative symptoms (eg, blunted affect, emotional withdrawal); and 16 assess general psychopathology (eg, poor attention, active social avoidance). Each item is scored on a 7-point scale (1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, and 7 = extreme). The PANSS total score can range from 30 to 210. A higher score indicates worse symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 6
Population: Intent-to-treat population: All participants who took at least 1 dose of double-blind investigational product and who had at least 1 post-baseline assessment of the primary efficacy parameter, the PANSS total score.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Cariprazine 4.5 mg | Risperidone 4.0 mg
Number analyzed (Participants) | 148 | 140 | 140 | 145 | 138
Units on a scale
  Baseline | 97.3 (0.8) | 97.1 (0.8) | 97.2 (0.7) | 96.7 (0.8) | 98.1 (0.8)
  Change at Week 6 | -9.5 (1.6) | -17.3 (1.7) | -18.7 (1.8) | -20.2 (1.6) | -25.3 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1.5 mg; Test type: Superiority or Other; p = 0.0005, ANCOVA; The analysis of covariance (ANCOVA) included treatment group and study center as factors and the Baseline PANSS total score as the covariate; Least squares mean difference = -7.5, 95% CI 2-sided [-11.8 to -3.3]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -8.8, 95% CI 2-sided [-13.1 to -4.6]
Statistical Analysis 3: Comparison: Placebo vs Cariprazine 4.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -10.4, 95% CI 2-sided [-14.6 to -6.2]
Statistical Analysis 4: Comparison: Placebo vs Risperidone 4.0 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -15.0, 95% CI 2-sided [-19.4 to -10.8]

2. Secondary Outcome: Change From Baseline to Week 6 in the CGI-S Score
Description: The Clinical Global Impressions-Severity (CGI-S) scale is a 7-point scale that measures the overall severity of the illness compared with the severity of illness in other patients the Investigator has observed. The Investigator assesses the severity of the patient's illness as one of the following: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patients. The CGI-S score can range from 1 to 7. A higher score indicates more severe illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Cariprazine 4.5 mg | Risperidone 4.0 mg
Number analyzed (Participants) | 148 | 140 | 140 | 145 | 138
Units on a scale
  Baseline | 4.9 (0.1) | 4.7 (0.1) | 4.9 (0.1) | 4.8 (0.1) | 4.8 (0.1)
  Change at Week 6 | -0.6 (0.1) | -0.9 (0.1) | -1.1 (0.1) | -1.2 (0.1) | -1.4 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1.5 mg; Test type: Superiority or Other; p = 0.0040, ANCOVA; The analysis of covariance (ANCOVA) included treatment group and study center as factors and the Baseline CGI-S score as the covariate; Least squares mean difference = -0.4, 95% CI 2-sided [-0.6 to -0.1]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; [statistical method as in outcome 2, analysis 1]; Least squares mean difference = -0.5, 95% CI 2-sided [-0.7 to -0.2]
Statistical Analysis 3: Comparison: Placebo vs Cariprazine 4.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Least squares mean difference = -0.6, 95% CI 2-sided [-0.9 to -0.4]
Statistical Analysis 4: Comparison: Placebo vs Risperidone 4.0 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Least squares mean difference = -0.8, 95% CI 2-sided [-1.1 to -0.6]

ADVERSE EVENTS:
Description: Safety population: All randomized participants who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Cariprazine 4.5 mg | Risperidone 4.0 mg
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/145 | 0/146 | 0/147 | 0/140
Serious Adverse Events (participants affected / at risk) | 7/151 | 5/145 | 0/146 | 4/147 | 3/140
Other Adverse Events (participants affected / at risk) | 67/151 | 73/145 | 74/146 | 87/147 | 80/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Cariprazine 1.5 mg (N=145) | Cariprazine 3.0 mg (N=146) | Cariprazine 4.5 mg (N=147) | Risperidone 4.0 mg (N=140)
Schizophrenia (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Agitation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
HIV test positive (Investigations) | 0 | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Fear of needles (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Psychotic behaviour (Psychiatric disorders) | 3 | 1 | 0 | 0 | 0
Spinal compression fracture (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Cariprazine 1.5 mg (N=145) | Cariprazine 3.0 mg (N=146) | Cariprazine 4.5 mg (N=147) | Risperidone 4.0 mg (N=140)
Nausea (Gastrointestinal disorders) | 5 | 7 | 11 | 11 | 9
Constipation (Gastrointestinal disorders) | 6 | 14 | 9 | 8 | 13
Vomiting (Gastrointestinal disorders) | 5 | 4 | 9 | 8 | 4
Weight increased (Investigations) | 1 | 3 | 5 | 0 | 7
Extrapyramidal disorder (Nervous system disorders) | 9 | 17 | 14 | 19 | 21
Akathisia (Nervous system disorders) | 8 | 13 | 14 | 13 | 12
Headache (Nervous system disorders) | 17 | 17 | 11 | 12 | 13
Sedation (Nervous system disorders) | 6 | 8 | 7 | 12 | 16
Dizziness (Nervous system disorders) | 3 | 5 | 3 | 9 | 8
Tremor (Nervous system disorders) | 6 | 5 | 7 | 4 | 10
Insomnia (Psychiatric disorders) | 11 | 15 | 24 | 24 | 21
Schizophrenia (Psychiatric disorders) | 12 | 6 | 7 | 9 | 1
Anxiety (Psychiatric disorders) | 5 | 6 | 8 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.